CLINICAL TRIAL: NCT04283396
Title: Study for Clinical Epidemiology and Methods of Diagnosis and Treatment of Novel Coronavirus Pneumonia (NCP)
Brief Title: Study for Novel Coronavirus Pneumonia (NCP)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Yang Jin, Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: NCP01
Record Dates: First submitted 2020-02-13; First posted 2020-02-25 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Novel Coronavirus Pneumonia
MeSH Terms: interventions — Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

INTERVENTIONS:
Combination Product: systemic treatment — Oxygen therapy, antiviral therapy, antibiotics, hormones, globulin

SUMMARY:
To develop practical and effective clinical diagnosis and treatment schemes for the control of novel coronavirus pneumonia.

DETAILED DESCRIPTION:
By retrospectively analyzing the clinical epidemiological characteristics of the novel coronavirus pneumonia and the current diagnosis and treatment schemes, as well as in-depth analyzing the disease development process and outcome trends of NCP patients to develop practical and effective clinical diagnosis and treatment schemes and provide guarantee for the rapid control of the epidemic.

ELIGIBILITY:
Inclusion Criteria:

* Patients confirmed with novel coronavirus pneumonia. The Diagnostic criteria refer to "Pneumonitis Diagnosis and Treatment Scheme for Novel Coronavirus Infection (Trial Version 5)";

Exclusion Criteria:

* Physician judged the patient was not suitable for this clinical trial.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients confirmed with novel coronavirus pneumonia.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-02-21 (Actual); Primary Completion 2020-05-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
recovery | up to 24 weeks
  Number of patients recover from novel coronavirus pneumonia

CONTACTS AND LOCATIONS:
Locations (1):
- Union hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided